CLINICAL TRIAL: NCT03995732
Title: Efficacy and Safety Evaluation of Phosphatidyl Choline Cu/Zn Superoxide Dismutase (PC-SOD) for Injection in Reducing Myocardial Reperfusion Injury: a Multicenter, Randomized, Single-blind, Placebo-controlled Dose-finding Study
Brief Title: Efficacy and Safety Evaluation of PC-SOD for Injection in Reducing Myocardial Reperfusion Injury
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tide Pharmaceutical Co., Ltd (Industry)
Collaborators: Peking University First Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CY-RD101-2; GUSU18003 (Other: GUSU Group)
Record Dates: First submitted 2019-06-05; First posted 2019-06-24 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Myocardial Reperfusion Injury
MeSH Terms: conditions — Myocardial Reperfusion Injury

STUDY DESIGN:
Who Masked: Participant
Masking Description: Since the appearance of PC-SOD preparations cannot be identical to that of placebo, and treatment groups have different administration doses, the study will be conducted in a single-blind manner, where only subjects (and families) are blinded and do not know whether they are treated by PC-SOD or placebo before unblinding.
  Interpretation of cardiac MRI and ECG will also be conducted in a blinding manner. Images of all subjects will be evaluated blindly by researchers not directly involved in the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 40 mg treatment group (Experimental): PC-SOD 40 mg dissolved in 10 mL of 5% glucose injection and intravenously administrated before recanalization.
  Interventions: Drug: PC-SOD
- 80 mg treatment group (Experimental): PC-SOD 80 mg dissolved in 10 mL of 5% glucose injection and intravenously administrated before recanalization.
  Interventions: Drug: PC-SOD
- 160 mg treatment group (Experimental): PC-SOD 160 mg dissolved in 10 mL of 5% glucose injection and intravenously administrated before recanalization.
  Interventions: Drug: PC-SOD
- placebo control group (Placebo Comparator): placebo dissolved in 10 mL of 5% glucose injection and intravenously administrated before recanalization.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: PC-SOD — PC-SOD will be dissolved in 10 mL of 5% glucose injection and intravenously administrated before recanalization.
  Arms: 160 mg treatment group; 40 mg treatment group; 80 mg treatment group
Drug: placebo — Placebo will be dissolved in 10 mL of 5% glucose injection and intravenously administrated before recanalization.
  Arms: placebo control group

SUMMARY:
The current study aims to evaluate different doses of PC-SOD injections for efficacy and safety in comparison to placebo, in order to provide a basis for future clinical trials in terms of experimental design and dose selection.

DETAILED DESCRIPTION:
The study is a randomized, single-blind, multi-center, placebo-controlled trial to preliminarily evaluate the efficacy and safety of PC-SOD, and to provide a basis for dose selection in the next stage of study.

For each participant, the trial will be divided into the screening/treatment (screening and treatment conducted during the first visit, 0 d) and safety follow-up (1 - 30 d) stages.

The study will screen 120 eligible subjects. After successful screening, the subjects will be randomly assigned into four groups of equal size, including the 40 mg PC-SOD, 80 mg PC-SOD, 160 mg PC-SOD and placebo control groups. Subjects in each group will be administered the corresponding intervention, followed by PCI treatment. During the safety follow-up stage, the subjects will receive basic treatment based on Guidelines for Management of Patients with ST-segment elevation myocardial infarction. Treatments will include dual anti-platelet therapy, beta-blockers, ACEI/ARB (angiotensin-converting enzyme inhibitor/ angiotensin receptor blocker), statins, anticoagulants, and so on.

By comparing the efficacy and safety endpoints of patients in the experimental and placebo control groups, the study aims to preliminarily evaluate the efficacy and safety of different doses of PC-SOD in reducing myocardial reperfusion injury.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 75 years, male or female;
2. Meeting the diagnostic criteria of AMI (chest pain for over 10 - 20 min, which could not be relieved completely by oral nitroglycerin; ST elevation ≥ 2 mm in two or more adjacent leads in leads V1-V5 );
3. Killip classes I or II;
4. Coronary angiography possible within 6 hours of onset;
5. Emergent coronary angiography showing occlusion in left anterior descending artery (TIMI grade 0 - 1); patients with this symptom could also be included despite inconformity to criterion 2);
6. Willingness to participate in the trial with ethical approval and informed consent provision.

Exclusion Criteria:

General exclusion criteria

1. Previous history of myocardial infarction;
2. History of myocardial revascularization before screening;
3. Thrombolytic treatment after onset;
4. Cardiogenic shock;
5. Cardiopulmonary resuscitation between onset and screening;
6. Atrial fibrillation, atrioventricular block (degree I, II or III), and other severe arrhythmias that cannot be corrected and affect hemodynamics;
7. Suspected of aortic dissection;
8. Diabetes with long-term insulin use, or definite macrovascular or small vascular lesions (stroke, diabetic nephropathy, retinopathy, diabetic foot, and etc.);
9. History of major surgeries within 6 months;
10. History of stroke within 6 months;
11. History of immune disorders within 6 months (such as cancer, lymphoma, HIV or hepatitis), or use of immunosuppressive agents at doses that can cause immunosuppression within 10 days;
12. Clinically significant diseases of the respiratory, digestive, blood, immune, endocrine, nervous or urinary systems (renal insufficiency in particular), and diseases that might cause serious risk to patients based on the judgement of researchers;
13. Allergy to two or more drugs and/or foods, or known allergy to sucrose;
14. Any contraindications for cardiac MRI, such as implantation of metal objects (pacemakers and/or implantable defibrillators; insulin pumps, or any other electronic devices; cerebral clips, aneurysm clips, and etc.), and other contraindications (such as claustrophobia);
15. Pregnancy or lactation in women;
16. Participation in other clinical trials within 3 months;
17. Situations considered unsuitable for enrollment (such as disease condition or patient compliance).

Exclusion criteria for angiography

1. Occlusion of left main artery;
2. Apart from the left anterior descending branch, other blood vessels requiring revascularization in the same period or within a month.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-06-18 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
The myocardial salvage index at 7 d after PCI | 7 days
  The myocardial salvage index is defined as (area of myocardial edema - area of myocardial infarction)/area of myocardial edema.
The area of myocardial infarction at 7 d after PCI (detected by delayed-enhanced MRI [Magnetic Resonance Imaging] ) | 7 days
  The area of myocardial infarction is defined as the percentage of left ventricular myocardium occupied by delayed enhancement.
Area of microvascular occlusion at 7 d after PCI | 7 days
  Microvascular occlusion is defined as the area with no enhancement in the infarcted regions where delayed enhancement can be observed on MRI scans.
The area of infarction determined by the AUC (area under curve) for CK-MB (creatine kinase-muscle/brain) at 72h after PCI. | 72 hours
  The area of infarction at 72h after surgery will be roughly estimated by calculating the AUC for CK-MB (before operation, and at 6, 12, 24, 48 and 72h after operation, respectively).
Cardiac function at 7 d after PCI | 7 days
  Cardiac function is assessed by assessing the left ventricular ejection fraction (percentage of stroke output to end-diastolic volume).
The TIMI (thrombolysis in myocardial infarction) grade of coronary blood flow after PCI. | within 24 hours
  Coronary artery reperfusion will be assessed by the TIMI grading system, whose grades include:
  Grade 0: no contrast filling at the occlusion site and distal end; Grade 1: the contrast passes some of the occluded sites, but cannot fill the distal vessels; Grade 2: the contrast can fill the distal end of coronary artery completely, but the filling and clearing of contrast is slower than that of normal coronary artery; Grade 3: the contrast can fill the distal end rapidly and completely, and can be removed quickly.
  The TIMI flow grades will be determined by two physicians separately. In case of disagreement, a lead physician will help make the final call.
The corrected TIMI frame count (cTFC) after PCI. | within 24 hours
  The left anterior descending (LAD) artery will be analyzed in a 30º right anterior oblique view with 30º cranial angulation. The left circumflex (LCX) will be analyzed in a 30º right anterior oblique view with 30º caudal angulation. The right coronary artery (RCA) will be analyzed in a 45º left anterior oblique view.
TIMI myocardial perfusion grade (TMPG) after PCI | within 24 hours
  Grade 0: no contrast entering the myocardium; Grade 1: the contrast enters myocardium slowly, with myocardial staining not disappearing or lasting for more than 30 s in the targeted vessels; Grade 2: delayed entering and disappearing of contrast in the myocardium, exceeding 3 cardiac cycles; Grade 3: normal entering and disappearing of contrast in the myocardium, occurring within 3 cardiac cycles.
Percentage of ST-segment resolution on ECG (electrocardiogram) at 90 min after PCI | 90 minutes
  ST-resolution is defined as more than 50% of resolution.
Number of cardiovascular events within 30 d after PCI | 30 days
  Cardiovascular events included all-cause death, cardiovascular death, non-fatal myocardial infarction, non-fatal stroke, and hospitalization due to heart failure.
SOD (Superoxide Dismutase) activity | 0 hours, 6 hours, 12 hours, 24 hours, 48 hours, 72 hours and 7 days after surgery
  Change from Baseline SOD activity at 6h, 12h, 24h, 48h, 72h and 7 d after surgery.
Occurence of adverse events | During patient hospitalization, up to 30 days
  Occurence of adverse events
Cardiac function at 30 d after PCI | 30 days
  Cardiac function is assessed by assessing the left ventricular ejection fraction (percentage of stroke output to end-diastolic volume).

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Wuhan Asia Heart Hospital, Wuhan, Hubei
  - Zhongshan Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yellon DM, Hausenloy DJ. Myocardial reperfusion injury. N Engl J Med. 2007 Sep 13;357(11):1121-35. doi: 10.1056/NEJMra071667. No abstract available. PMID 17855673
- [Background] Zweier JL. Measurement of superoxide-derived free radicals in the reperfused heart. Evidence for a free radical mechanism of reperfusion injury. J Biol Chem. 1988 Jan 25;263(3):1353-7. PMID 2826476
- [Background] Werns SW, Lucchesi BR. Free radicals and ischemic tissue injury. Trends Pharmacol Sci. 1990 Apr;11(4):161-6. doi: 10.1016/0165-6147(90)90068-J. PMID 2185587
- [Background] Kloner RA, Przyklenk K, Whittaker P. Deleterious effects of oxygen radicals in ischemia/reperfusion. Resolved and unresolved issues. Circulation. 1989 Nov;80(5):1115-27. doi: 10.1161/01.cir.80.5.1115. PMID 2553296
- [Background] Przyklenk K, Kloner RA. Superoxide dismutase plus catalase improve contractile function in the canine model of the "stunned myocardium". Circ Res. 1986 Jan;58(1):148-56. doi: 10.1161/01.res.58.1.148. PMID 3943152
- [Background] Engler R, Gilpin E. Can superoxide dismutase alter myocardial infarct size? Circulation. 1989 May;79(5):1137-42. doi: 10.1161/01.cir.79.5.1137. No abstract available. PMID 2653661
- [Background] Igarashi R, Hoshino J, Ochiai A, Morizawa Y, Mizushima Y. Lecithinized superoxide dismutase enhances its pharmacologic potency by increasing its cell membrane affinity. J Pharmacol Exp Ther. 1994 Dec;271(3):1672-7. PMID 7996483
- [Background] Wu E, Ortiz JT, Tejedor P, Lee DC, Bucciarelli-Ducci C, Kansal P, Carr JC, Holly TA, Lloyd-Jones D, Klocke FJ, Bonow RO. Infarct size by contrast enhanced cardiac magnetic resonance is a stronger predictor of outcomes than left ventricular ejection fraction or end-systolic volume index: prospective cohort study. Heart. 2008 Jun;94(6):730-6. doi: 10.1136/hrt.2007.122622. Epub 2007 Dec 10. PMID 18070953